CLINICAL TRIAL: NCT00533676
Title: A Randomized, Double-Blind, Placebo-Controlled Endpoint Selection and Questionnaire Validation Study to Assess the Niacin Induced Flushing Caused by NIASPAN (TM)
Brief Title: Endpoint Validation Study (0524A-015)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-015; MK0524A-015; 2007_612
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Flushing
MeSH Terms: conditions — Flushing | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0524A, /Duration of Treatment : 8 Weeks
Drug: Comparator : placebo (unspecified) /Duration of Treatment : 8 Weeks

SUMMARY:
To determine the most effective daily dose of MK0524A when compared with placebo after the 8-week treatment period for Niacin Induce Flushing (NIF).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female between 18 to 70 years
* Qualified women must be sterile (through surgery) and/or post-menopausal, and/or agree to use birth control

Exclusion Criteria:

* You are a woman who is having hot flashes, receiving Hormone Replacement Therapy (HRT), and/or other therapies for hot flashes
* You are currently using Niacin/or Niacin containing products with a daily dose over 50 mg/day
* You are sensitive to niacin
* You have a history gout
* You drink more than 2 glasses of alcohol per day and you are not willing to stop
* You don't have access to a telephone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the most effective daily dose and measurements to assess acute and chronic (long-lasting) Niacin Induce Flushing (NIF). | 8 weeks

SECONDARY OUTCOMES:
To assess the the time points of Niacin Induce Flushing (NIF) across the 8-week treatment period. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Norquist JM, Watson DJ, Yu Q, Paolini JF, McQuarrie K, Santanello NC. Validation of a questionnaire to assess niacin-induced cutaneous flushing. Curr Med Res Opin. 2007 Jul;23(7):1549-60. doi: 10.1185/030079907x199637. PMID 17559750
- [Background] Paolini JF, Mitchel YB, Reyes R, Thompson-Bell S, Yu Q, Lai E, Watson DJ, Norquist JM, Sisk CM, Bays HE. Measuring flushing symptoms with extended-release niacin using the flushing symptom questionnaire: results from a randomised placebo-controlled clinical trial. Int J Clin Pract. 2008 Jun;62(6):896-904. doi: 10.1111/j.1742-1241.2008.01739.x. Epub 2008 Apr 10. PMID 18410350
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/policies-perspectives.html